CLINICAL TRIAL: NCT05113134
Title: A Prospective Clinical Study of Transvaginal Versus Transabdominal Extraction of Laparoscopically-excised Specimen (STTELS)
Brief Title: Transvaginal Versus Transabdominal Extraction of Laparoscopically-excised Specimen
Acronym: STTELS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUBH B-1411-276-005
Record Dates: First submitted 2021-11-05; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Colorectal Neoplasms; Urologic Neoplasms; Gastrointestinal Neoplasms; Neoplasms by Site
Keywords: natural orifice specimen extraction; laparoscopic surgery; transvaginal; Female
MeSH Terms: conditions — Colorectal Neoplasms; Urologic Neoplasms; Gastrointestinal Neoplasms; Neoplasms by Site

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transvaginal natural orifice specimen extraction (NOSE) (Experimental): The outcomes of transvaginal natural orifice specimen extraction (NOSE) in patients who underwent multiport laparoscopic surgery for resection of solid organs including kidney, liver, stomach, adrenal gland and bladder
  Interventions: Procedure: Transvaginal natural orifice specimen extraction (NOSE)

INTERVENTIONS:
Procedure: Transvaginal natural orifice specimen extraction (NOSE) — Under general anesthesia, patients who are planned to perform multiport laparoscopic surgery for resection of solid organs including kidney, liver, stomach, adrenal gland and bladder will undergo Transvaginal NOSE

SUMMARY:
The aim of this study is to evaluate the outcomes of transvaginal natural orifice specimen extraction (NOSE) in patients who are planning multiport laparoscopic surgery for resection of solid organs including kidney, liver, stomach, adrenal gland and bladder.

DETAILED DESCRIPTION:
Study design:

This was a prospective, single center, single arm study. This clinical trial was approved by the Institutional Review Boards.

Study process:

All patients gave informed written consent after being informed of the details of the study. All participants underwent demographic and history taking, laboratory tests and a gynecological examination to determine whether specimen removal through vagina is possible. The patients who was adequate for this study were planned to perform multiport laparoscopic surgery and patients were subjected to transvaginal NOSE.

To perform transvaginal NOSE procedure, the patients were placed in the lithotomy position with Trendelenburg position. After about 1-2cm incision at the posterior vaginal fornix, endopouch was introduced into the abdominal cavity through vaginal incision site. The specimen was placed inside a endopouch and removed through vagina. Closure of vaginal incision site was achieved by transvaginally with 2/0 absorbable suture.

During the second and third visit at 1 week and 8 week, Patient and Observer Scar Assessment Scale (POSAS) was performed to assess cosmetic outcomes of scar. Subjects with sexual activity carried out Female Sexual Function Index (FSFI) questionnaire to assess sexual function at final visit which occurred at 6 months after surgery.

Statistical analysis:

All data are summarized as means ± standard deviation or as numbers with proportions. A p < 0.05 was considered to indicate significance. Student's t-test and Mann-Whitney U test were conducted to compare continuous parametric variables and non-parametric variables, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are accessible with vaginal approach
* Patients scheduled for laparoscopic resection of stomach, colon, kidney and spleen for benign or malignant diseases
* Patients with normal cervical cancer screening tests within the last 3 years except inflammatory findings

Exclusion Criteria:

* Patients without sexual intercourse
* Patients who are considered unable to remove specimen through vagina due to narrow introitus in gynecological examination
* Patients who are expected to have severe adhesion due to deep infiltrative endometriosis or previous pelvic surgery history
* Patients with abnormal cervical cancer screening tests
* Patients scheduled to perform concomitant hysterectomy

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
Patient and Observer Scar Assessment Scale (POSAS) | 8 week
  Cosmetic outcomes of scar assessed by Patient and Observer Scar Assessment Scale (POSAS) 1 week and 8 weeks after surgery. The POSAS is the international validated scar assessment questionnaire that measures quality of the scar from the perspective of both patient and observer.

SECONDARY OUTCOMES:
Female Sexual Function Index (FSFI) questionnaire | 6 months
  Sexual function assessment

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Soyman Z, Kelekci S, Aydogmus S, Demirel E, Ekmekci E. Transabdominal versus transvaginal specimen extraction in mini-laparoscopic surgery. J Obstet Gynaecol Res. 2019 Dec;45(12):2400-2406. doi: 10.1111/jog.14134. Epub 2019 Oct 3. PMID 31580003
- [Result] Park JS, Kang H, Park SY, Kim HJ, Lee IT, Choi GS. Long-term outcomes after Natural Orifice Specimen Extraction versus conventional laparoscopy-assisted surgery for rectal cancer: a matched case-control study. Ann Surg Treat Res. 2018 Jan;94(1):26-35. doi: 10.4174/astr.2018.94.1.26. Epub 2017 Dec 28. PMID 29333423
- [Result] Guan X, Liu Z, Longo A, Cai JC, Tzu-Liang Chen W, Chen LC, Chun HK, Manuel da Costa Pereira J, Efetov S, Escalante R, He QS, Hu JH, Kayaalp C, Kim SH, Khan JS, Kuo LJ, Nishimura A, Nogueira F, Okuda J, Saklani A, Shafik AA, Shen MY, Son JT, Song JM, Sun DH, Uehara K, Wang GY, Wei Y, Xiong ZG, Yao HL, Yu G, Yu SJ, Zhou HT, Lee SH, Tsarkov PV, Fu CG, Wang XS; International Alliance of NOSES. International consensus on natural orifice specimen extraction surgery (NOSES) for colorectal cancer. Gastroenterol Rep (Oxf). 2019 Feb;7(1):24-31. doi: 10.1093/gastro/goy055. Epub 2019 Jan 23. PMID 30792863
- [Derived] Hwang WY, Suh DH, Lee S. Cosmesis and feasibility of transvaginal natural orifice Specimen extraction (NOSE) for large organ specimen: a prospective pilot study. BMC Urol. 2022 Oct 29;22(1):165. doi: 10.1186/s12894-022-01114-4. PMID 36309743